CLINICAL TRIAL: NCT03130426
Title: Remission Evaluation of a Metabolic Intervention for Type 2 Diabetes With IGlarLixi
Acronym: REMIT-iGL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIT-iGlarLixi
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; iGlarLixi; Metformin; Insulin; Diet; Exercise; Lifestyle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Motor Activity | interventions — Insulin Glargine; lixisenatide; Metformin; Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Drug: iGlarLixi - sc injection; Drug: metformin - oral administration; Drug: insulin glargine - sc injection; Behavioral: lifestyle therapy, diet and exercise
  Interventions: Drug: iGlarLixi; Drug: Insulin Glargine; Drug: Metformin; Behavioral: Lifestyle therapy
- Standard Care (No Intervention): Standard glycemic care as informed by the current clinical practice guidelines

INTERVENTIONS:
Drug: iGlarLixi — Dose is titrated to achieve fasting normoglycemia
  Other Names: glargine insulin / lixisenatide
  Arms: Intervention
Drug: Insulin Glargine — In those who need additional insulin or who cannot tolerate iGlarLixi, insulin glargine will be used. Dose is titrated to achieve fasting normoglycemia.
  Other Names: Lantus
  Arms: Intervention
Drug: Metformin — Dose is titrated to 2000 mg daily or maximal tolerated dose
  Arms: Intervention
Behavioral: Lifestyle therapy — Lifestyle intervention includes individualized dietary and exercise advice and frequent visits for goal reinforcement, behavior modification and problem-solving
  Other Names: diet and exercise
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine whether in patients with early type 2 diabetes, a short-term intensive metabolic intervention comprising iGlarLixi, metformin, and lifestyle approaches will be superior to standard diabetes therapy in achieving sustained diabetes remission.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized controlled trial in 160 patients with recently-diagnosed T2DM. Participants will be randomized to 2 treatment groups: (a) a 12-week course of treatment with iGlarLixi, metformin and lifestyle therapy, and (b) standard diabetes therapy, and followed for a total of 64 weeks (1 year and 3 months). In all participants with HbA1C<7.3% at the 12 week visit, glucose-lowering medications will be discontinued and participants will be encouraged to continue with lifestyle modifications and regular glucose monitoring. Participants with HbA1C ≥ 7.3% at this visit or who experience hyperglycemia relapse after stopping drugs will receive standard glycemic management as informed by the current Canadian Diabetes Association clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged 30-80 years;
2. type 2 diabetes mellitus within 5 years of diagnosis;
3. stable diabetes drug regimen in the 10 weeks before randomization;
4. HbA1c 6.5-9.5% on no glucose lowering drugs, or </= 8.5% on 1 glucose-lowering drug, or </= 8.0% on 2 glucose lowering drugs;
5. body mass index >/= 23 kg/m2;
6. ability and willingness to perform self-monitoring of capillary blood glucose (SMBG);
7. ability and willingness to self-inject iglarlixi; and
8. provision of informed consent.

Exclusion Criteria:

1. current use of insulin therapy;
2. history of hypoglycemia unawareness, or severe hypoglycemia requiring assistance;
3. history of end-stage renal disease or renal dysfunction as evidenced by eGFR<45 mL/min/1.73 m2 by MDRD formula;
4. history of lactic acidosis or diabetic ketoacidosis;
5. active liver disease or elevated alanine transferase (ALT) levels >\= 2.5 times upper limit of normal at the time of enrolment;
6. history or clinical suspicion of pancreatitis or medullary thyroid cancer, or a calcitonin level >/= 20 pg/ml;
7. cardiovascular disease (unless cleared for a moderate intensity exercise program by a specialist) including: i. acute coronary syndrome, hospitalization for unstable angina, myocardial infarction, or revascularization with coronary artery bypass grafting or percutaneous coronary intervention; ii. peripheral vascular disease, valvular heart disease, cardiomyopathy, aortic dissection, tachyarrhythmias, bradyarrhythmias, prior stroke or TIA; iii. prior hospitalization for heart failure; or iv. ECG findings concerning for ischemic heart disease (i.e. pathological Q-waves, ST-segment-T-wave abnormalities in contiguous leads, left anterior hemiblock, left bundle branch block, second or third degree atrioventricular block).
8. history of any disease requiring frequent intermittent or continuous systemic glucocorticoid treatment;
9. history of bariatric surgery, or planned bariatric surgery in the next 1.5 years;
10. history of any major illness with a life expectancy of < 3 years;
11. history of injury or any other condition that significantly limits participant's ability to achieve moderate levels of physical activity;
12. excessive alcohol intake, acute or chronic;
13. currently pregnant, or breastfeeding, or not using a reliable method of birth control for the duration of the trial in all females with childbearing potential;
14. inability to take glargine, lixisenatide or metformin

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The first occurrence of diabetes relapse | 64 weeks of follow-up

SECONDARY OUTCOMES:
Number of participants achieving drug-free diabetes remission | 24 weeks after randomization
  Diabetes remission is defined as HbA1C < 6.5% off diabetes drugs for at least 12 weeks
Number of participants achieving drug-free normoglycemia defined as HbA1C < 6.0% off diabetes drugs for at least 12 weeks | 24 weeks after randomization
Percentage of weight loss from baseline | 12 weeks
  (Weight at randomization - weight at 12 weeks)/(weight at randomization)
Change in waist circumference from baseline | 12 weeks
  (Waist circumference at 12 weeks - weight circumference at randomization)
Glycated hemoglobin (HbA1C) | 12 weeks
  Expressed in Diabetes Control and Complications Trial (DCCT) units

CONTACTS AND LOCATIONS:
Overall Officials: Natalia McInnes, MD, Principal Investigator — McMaster University; Hertzel Gerstein, MD, Principal Investigator — McMaster University
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - LMC, Burlington, Ontario
  - Joanne Liutkus, Cambridge, Ontario
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Western University, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No